CLINICAL TRIAL: NCT03493789
Title: A Pilot Study of FDG-PET Variability to Establish Biology-Guided Treatment Planning Feasibility for Stereotactic Body Radiation Therapy
Brief Title: Fludeoxyglucose F-18-PET in Planning Lung Cancer Radiation Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: RefleXion Medical (Industry); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kristin Higgins, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00101066; NCI-2018-00375 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD4267-17 (Other: Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2018-03-20; First posted 2018-04-11 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Stage I Lung Cancer; Stage I Non-Small Cell Lung Cancer AJCC v7; Stage IA Non-Small Cell Lung Carcinoma AJCC v7; Stage IB Non-Small Cell Lung Carcinoma AJCC v7; Stage II Lung Cancer; Stage II Non-Small Cell Lung Cancer AJCC v7; Stage IIA Non-Small Cell Lung Carcinoma AJCC v7; Stage IIB Non-Small Cell Lung Carcinoma AJCC v7
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (FDG-PET, SBRT) (Experimental): Participants receive fludeoxyglucose F-18 IV and after 60 minutes undergo positron emission tomography (PET) within 4 weeks of the first planned stereotactic body radiation therapy (SBRT) fraction, prior to the second planned fraction, and prior to the fifth planned fraction.
  Interventions: Drug: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography (PET); Radiation: Stereotactic Body Radiation Therapy (SBRT)

INTERVENTIONS:
Drug: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose
Procedure: Positron Emission Tomography (PET) — Undergo FDG-PET
  Other Names: Medical imaging, positron emission tomography; PET scan; Positron emission tomography scan; Proton magnetic resonance spectroscopic imaging
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Undergo SBRT
  Other Names: SABR; Stereotactic ablative body radiation therapy

SUMMARY:
This trial studies how well fludeoxyglucose F-18 - positron emission tomography (PET) works in planning radiation therapy in participants with early non-small cell lung cancer, early stage lung cancer, or cancer that has spread to lungs from other parts of the body. Using PET in addition to the standard computed tomography to plan radiation therapy for cancer may help doctors to maximize the dose to the cancer and minimize the dose to normal tissues.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To determine the maximum inter-fraction variability of fludeoxyglucose F-18 (18-F FDG)-PET activity of thoracic tumor treatment volumes through a 5-fraction stereotactic body radiation therapy (SBRT) course as it relates to the planning feasibility of emission-guided radiation therapy, or biologically-guided radiation therapy (BgRT).

SECONDARY OBJECTIVES:

I. To compare similar inter-fraction variability of FDG-PET activity for non-thoracic SBRT target volumes for the purpose of determining the feasibility of BgRT.

II. To compare dosimetric endpoints for primary tumor coverage and dose to organs at risk between conventional SBRT planning and simulated BgRT, or emission-guided radiation therapy planning for thoracic and non-thoracic targets.

III. To compare dosimetry for primary tumor coverage and dose to organs at risk between adaptive cone beam computed tomography (CT) planning, and simulated adaptive emission-guided radiation therapy (BgRT) planning for thoracic and non-thoracic targets.

IV. To compare variability of 18-F FDG-PET in patients undergoing immunotherapy simultaneously during SBRT, or within 4 weeks of SBRT treatment with patients undergoing SBRT but not receiving immunotherapy.

OUTLINE:

Participants receive fludeoxyglucose F-18 intravenously (IV) and after 60 minutes undergo PET within 4 weeks of the first planned SBRT fraction, prior to the second planned fraction, and prior to the fifth planned fraction.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are offered radiotherapy using a 5-fraction stereotactic body radiation therapy course, at the recommendation of the treating radiation oncologist
* Patients with early non-small cell lung carcinoma, or clinically-diagnosed early stage lung cancer, or pulmonary metastases
* Patients with a limited (1-5) number of metastatic foci outside of the thorax who are candidates for consolidative treatment with SBRT
* Patient with either a single focus or multiple foci (multi-isocentric planning) of disease in the thorax amenable to SBRT with at least one focus with at least 1.5 cm or larger in its largest diameter
* Patients who are planned to receive either chemotherapy, targeted therapy, immunotherapy, or no additional cancer-directed drug therapy

Exclusion Criteria:

* Prior radiation therapy which would provide significant dose overlap with the planned target volume(s) delivered within 30 days of enrollment or registration
* Major invasive surgical procedure occurring between the first treatment-eligible PET/CT examination and end of radiotherapy that would affect the treatment target region
* Patients with minimal FDG-avidity localized to the planned treatment target (e.g. maximum standardized uptake value [SUV] < 4.0)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Change in metabolic tumor volumes measuring inter-fraction variability of fludeoxyglucose F-18-PET (FDG) - positron emission tomography (PET) activity of thoracic stereotactic body radiation therapy (SBRT) target volumes | Up to 6 weeks from study start
  Metabolic tumor volumes across the treatment continuum, i.e. pre-treatment, before second fraction and before the last fraction of treatment, will be compared. The observed % change from baseline will be calculated at all time points for all 15 patients and for every tumor treated with SBRT.
Change in total lesion glycolysis values measuring inter-fraction variability of fludeoxyglucose F-18-PET (FDG) - positron emission tomography (PET) activity of thoracic stereotactic body radiation therapy (SBRT) target volumes | Up to 6 weeks from study start
  Total lesion glycolysis values across the treatment continuum, i.e. pre-treatment, before second fraction and before the last fraction of treatment, will be compared. The observed % change from baseline will be calculated at all time points for all 15 patients and for every tumor treated with SBRT.

SECONDARY OUTCOMES:
Change in metabolic tumor volumes measuring inter-fraction variability of fludeoxyglucose F-18-PET (FDG) - positron emission tomography (PET) activity of non-thoracic stereotactic body radiation therapy (SBRT) target volumes | Up to 6 weeks from study start
  Metabolic tumor volumes across the treatment continuum, i.e. pre-treatment, before second fraction and before the last fraction of treatment, will be compared. The observed % change from baseline will be calculated at all time points for all 15 patients.
Change in total lesion glycolysis values measuring inter-fraction variability of fludeoxyglucose F-18-PET (FDG) - positron emission tomography (PET) activity of non-thoracic stereotactic body radiation therapy (SBRT) target volumes | Up to 6 weeks from study start
  Total lesion glycolysis values across the treatment continuum, i.e. pre-treatment, before second fraction and before the last fraction of treatment, will be compared. The observed % change from baseline will be calculated at all time points for all 15 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Higgins, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States

DOCUMENTS (1):
  • Informed Consent Form (2018-11-05): https://cdn.clinicaltrials.gov/large-docs/89/NCT03493789/ICF_000.pdf